CLINICAL TRIAL: NCT05176067
Title: Department of Thoracic Oncology, Affiliated Tumor Hospital of Guizhou Medical University
Brief Title: Randomized Controlled Clinical Study of Drug Therapy Combined With Thoracic Radiotherapy for Non-oligometastatic NSCLC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guizhou Medical University (Other)
Responsible Party: Principal Investigator, Bing Lu, Chief physician, Guizhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Guizhou MU
Record Dates: First submitted 2021-11-27; First posted 2022-01-04 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Clinical Study
Who Masked: Investigator
Masking Description: Randomized Controlled Clinical Study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- drug therapy group (No Intervention): targeted therapy, immune, chemotherapy
- drug therapy concurrent radiotherapy (Experimental): drug therapy(targeted therapy, immune, chemotherapy ) combined with thoracic tumor concurrent radiotherapy
  Interventions: Radiation: Thoracic Three-dimensional Radiotherapy

INTERVENTIONS:
Radiation: Thoracic Three-dimensional Radiotherapy — Drug Therapy Combined With Thoracic Three-dimensional Radiotherapy
  Arms: drug therapy concurrent radiotherapy

SUMMARY:
To investigate whether radiotherapy combined with drug therapy is beneficial to non- oligometastatic stage IV NSCLC

DETAILED DESCRIPTION:
Group A (targeted therapy, immunotherapy, chemotherapy); The efficacy was evaluated after the second and fourth cycles of chemotherapy and immunotherapy; The efficacy of targeted therapy was evaluated every month; Group B (drug concurrent radiotherapy group: combined with thoracic primary tumor radiotherapy on the basis of targeted therapy, immune, chemotherapy ) The efficacy was evaluated after the second and fourth cycles of chemotherapy and immunotherapy; The efficacy of targeted therapy was evaluated every month; Radiographic evaluation was performed after radiotherapy for the primary lesion of the chest.

ELIGIBILITY:
Inclusion Criteria:

1. Non- small cell lung cancer patients diagnosed by pathology or cytology;
2. Patients with stage IV non-oligometastasitatic [Eighth Edition];
3. initial treatment (no previous treatment);
4. age 18 ~ 80 years old, physical condition score ECOG 0 ~ 2 or KPS ≥ 60;
5. distance metastatic lesions: more than 5 metastatic lesions ; mind when brain metastases; The number of pulmonary metastases does not affect lung function, and radiotherapy for primary and/or partial metastases may be performed;
6. no contraindications such as radiotherapy, EGFR-TKI, chemotherapy, and immunotherapy;
7. primary tumor radiotherapy requires IMRT technology; In the plan design, the primary tumor prescription dose (DTGTV) was given under the damage control threshold standard, and the prescription dose was ≥ 40Gy; During the planned evaluation, the prescription dose includes 100% GTV, and 90% prescription dose includes 98% ~ 100% PTV [planned target dose (DTP) ≥ 36Gy]; Normal lung (whole lung volume minus GTV volume) V20 ≤ 32%, MLD ≤ 20GY; (V20 ≤ 25% in radiotherapy for patients with ALK, Ros-1, met, etc.).
8. radiotherapy for metastatic tumors is three-dimensional radiotherapy technology (IMRT / SRT / SBRT / VMAT, etc.), SBRT.
9. the subject has no dysfunction of main organs, or the laboratory test indicators must meet the following requirements: hematology: it is within the normal range according to the standards of each laboratory; Cardiac function: normal range; Liver function: normal range; Renal function: normal range; Pulmonary function: FEV1 > 50%, mild to moderate impairment of pulmonary function.
10. The sign informed consent before treatment (radiotherapy, chemotherapy, immunization, targeted drug therapy);
11. patients have good compliance with the treatment and follow-up.

Exclusion Criteria:

1. Patients with pathological type, stage, and survival status that do not meet the inclusion criteria;
2. Stage IV NSCLC patients with serous effusion such as malignant pleural effusion and pericardial effusion;
3. Patients with extensive liver metastasis and intrapulmonary metastasis have seriously affected liver and lung function;
4. The patient had no control of hypertension, diabetes, unstable angina, history of myocardial infarction, or had congestive heart failure or cardiac arrhythmia in the past 12 months. Heart valve disease with definite clinical diagnosis; Disease activity period of bacterial, fungal, or viral infection; Mental disorders; Severe impairment of pulmonary function;
5. Pregnant and lactating patients;
6. Patients with a history of other active malignant tumors except for small cell lung cancer before enrollment; Non-melanoma skin basal cell carcinoma, cervical carcinoma in situ and cured early prostate cancer are excluded;
7. Patients with the allergic constitution and known or suspected allergy to any drug in the study without alternative drugs;
8. Patients with poor compliance;
9. The researcher believes that it is not suitable to participate in this experiment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2021-12-30 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | through study completion, an average of 1 year
  The PFS of primary lung lesions and mediastinal metastatic lymph nodes
ORR | through study completion, an average of 1-2 years
  evaluate efficacy of drug therapy，efficacy of drug combination with radiotherapy with RECIST criteria.

SECONDARY OUTCOMES:
Toxicity and side effecttion | through study completion, an average of 1-2 years
  CTC5.0 standard was used to evaluate toxicity and side effects caused by drug therapy and radiotherapy.such as Pulmonary toxicity,Hematological toxicity,esophagitis.

CONTACTS AND LOCATIONS:
Overall Officials: Bing Lu, bachelor, Study Chair — Department of thoracic oncology, Affiliated Cancer Hospital of Guizhou Medical University

IPD SHARING:
Plan to Share IPD: No